CLINICAL TRIAL: NCT07112677
Title: Seroprevalence of Brucella Antibodies in High-Risk Patients With Low Back Pain: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Elham Ahmed Hassan (Other)
Responsible Party: Sponsor-Investigator, Elham Ahmed Hassan, Professor of Tropical Medicine and Gastroenterology, Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AUN-BRU-LBP-2024
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Brucellosis; Low Back Pain
Keywords: brucella antibodies; low back pain
MeSH Terms: conditions — Brucellosis; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1 (Patients): Low Back Pain Group, Group 2 (Controls): Control Group
  Interventions: Diagnostic Test: Brucella Antibody Testing (ELISA)

INTERVENTIONS:
Diagnostic Test: Brucella Antibody Testing (ELISA) — Serological testing for Brucella antibodies using the SERION ELISA classic Brucella IgG/IgM/IgA kit (Institut Virion\Serion GmbH, Würzburg, Germany). The test detects Brucella-specific IgG, IgM, and IgA antibodies in serum samples to assess current or past exposure. All samples were processed and interpreted according to the manufacturer's instructions. This diagnostic intervention was used for both the low back pain group and the control group.

SUMMARY:
The goal of this observational case-control study is to assess the presence of Brucella antibodies in patients with low back pain who are at high risk for brucellosis exposure, such as those with animal contact or consumption of unpasteurized dairy products. The main question it aims to answer is:

Is there a significant association between Brucella seropositivity and low back pain in high-risk individuals?

Researchers will compare patients with low back pain to age- and sex-matched healthy controls without back pain but with similar exposure risks, to see if Brucella antibodies are more frequent in the patient group.

Participants will:

Undergo a detailed clinical history and physical examination

Provide blood samples for serological testing using ELISA for Brucella IgG/IgM/IgA

Be evaluated for other symptoms such as fever, fatigue, and joint pain

ELIGIBILITY:
Inclusion Criteria:

* Adults of any sex at high risk of Brucella exposure (e.g., contact with livestock or consumption of unpasteurized dairy products)
* Patients presenting with non-specific low back pain
* Willing and able to provide informed consen

Exclusion Criteria:

* Evidence of tuberculosis (Pott's disease)
* Evidence of septic spondylitis
* Known metastatic bone lesions
* Known degenerative or autoimmune rheumatologic spinal diseases
* History of prior spinal surgery or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with high risk of Brucella exposure (e.g., animal contact or consumption of unpasteurized dairy products), including patients presenting with non-specific low back pain and healthy controls without back pain. Participants were recruited from outpatient clinics and inpatient wards at Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of Brucella Antibodies in High-Risk Patients with Low Back Pain | February 2024 to February 2025
  The presence of Brucella antibodies (IgG, IgM, and IgA) in serum was assessed using the SERION ELISA classic Brucella kit. A positive result indicates prior or current exposure to Brucella species. The outcome compares the proportion of seropositive individuals between patients with low back pain and matched controls.
Prevalence of Brucella Antibodies in High-Risk Patients with Low Back Pain | At enrollment
  The presence of Brucella antibodies (IgG, IgM, and IgA) in serum was assessed using the SERION ELISA classic Brucella kit. A positive result indicates prior or current exposure to Brucella species. The outcome compares the proportion of seropositive individuals between patients with low back pain and matched controls.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University Hospital, Asyut
  - Assiut University, Asyut

IPD SHARING:
Plan to Share IPD: No
I do not have specific consent from participants to share individual-level data.